CLINICAL TRIAL: NCT05366361
Title: The Dynamics of Human Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Stanford University
Other Study IDs: 57424
Record Dates: First submitted 2022-04-22; First posted 2022-05-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: ablation; arrhythmias, cardiac; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients Undergoing Clinically-Indicated Maze Surgery: This group includes patients with persistent AF who will be undergoing clinically-indicated Maze surgery.
- Patients Undergoing Clinically-Indicated Ablation: This groups includes patients with persistent AF who will be undergoing clinically-indicated ablation.

SUMMARY:
Atrial fibrillation (AF) is an enormous public health problem in the United States, affecting 2-5 million Americans and causing rapid heart beats, stroke, heart failure or death. In this project, the applicant will develop a novel framework to better understand human AF that builds on agreement between several concepts for the disease. The applicant will develop strategies to identify AF patients who will best respond to each of several therapies, to guide personalized therapy.

DETAILED DESCRIPTION:
The specific aim of this clinical study is to identify patients who will or will not respond to PVI, PVI plus other ablation or Maze surgery based on locations of organized-to-disorganized areas and clinical profile. We will develop non-invasive ECGI and intracardiac recordings in our registry, then test them prospectively in an observational study.

Premise: Identifying responders or non-responders to PVI alone, or PVI plus other ablation or Maze surgery may enable patient-tailored therapy. This may raise overall success, reduce risks from unsuccessful procedures and improve resource utilization(58,128-130). This proposal will prospectively test in single-arm observations studies if patients who exhibit large organized AF areas at planned ablation regions have higher procedural success than patients with smaller areas. We will use non-invasive ECGI indices of organized AF, based on Preliminary data(9, 84, 85).

This project is significant because it will establish a deeper understanding of AF and will develop strategies to identify AF patients who will best respond to each of several therapies, to guide personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* referred for ablation or Maze surgery at Stanford Medicine for persistent AF (i.e. which requires cardioversion to terminate and/or lasts >7 days)
* Per our clinical practice and guidelines (Calkins et al., Heart Rhythm 2018), patients will have failed or be intolerant of >or= 1 anti-arrhythmic drug. Patients after Maze surgery typically have failed prior endocardial ablation.

Exclusion Criteria:

* active coronary ischemia or decompensated heart failure
* atrial or ventricular clot on trans-esophageal echocardiography
* pregnancy (to minimize fluoroscopic exposure)
* inability or unwillingness to provide informed consent
* rheumatic valve disease (results in a unique AF phenotype)
* thrombotic disease or venous filters
* prior chest surgery is a relative contraindication for Maze surgery

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include men and women of any ethnicity aged >21 years referred for ablation or Maze surgery at Stanford Medicine for persistent AF (i.e. which requires cardioversion to terminate and/or lasts >7 days). Per our clinical practice and guidelines (Calkins et al., Heart Rhythm 2018), patients will have failed or be intolerant of >or= 1 anti-arrhythmic drug. Patients after Maze surgery typically have failed prior endocardial ablation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Does the Area of Organized Regions in AF predict success from Ablation? | 1 year.
  We will map areas of organized activity in all patients. We will compare if patients with success from ablation (absence of recurrent AF or atrial tachycardia on outpatient monitoring) have larger organized areas than those without success.

SECONDARY OUTCOMES:
Does ablation through larger organized areas explain success from ablation. | 1 year
  We will map areas of organized activity in all patients. We will compare if patients with ablation lesions through organized areas, or that eliminates organized areas, have higher or lower success from ablation (determined by absence of recurrent AF or atrial tachycardia on outpatient monitoring) than patients in whom ablation did not encroach on organized areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No